CLINICAL TRIAL: NCT03725982
Title: Work Physiological-Biomechanical Analysis of a Passive Exoskeleton to Support Occupational Lifting and Flexing Processes
Acronym: ADVANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Audi AG (Industry); BASF (Industry); BMW AG (Industry); Dachser Intelligent Logistics (Industry); Daimler AG (Industry); Deutsche Post AG (Industry); Iturri Gruppe (Industry); MTU Aero Engines AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UKT-2018-AS0-1836
Record Dates: First submitted 2018-09-27; First posted 2018-10-31 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2019-05

CONDITIONS: Passive Upper-limb Exoskeleton
Keywords: passive exoskeleton; forward trunk flexion; trunk rotation; muscle activity; inverse dynamics; modelling
MeSH Terms: interventions — Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: 1. Static sorting Six conditions as combination of exoskeleton (without vs. with) and trunk posture (forward flexion vs. flexion + rotation left vs. flexion + rotation right) are investigated in a randomized order.
  2. Dynamic lifting Twelve conditions as combination of exoskeleton (without vs. with), work posture (forward flexion vs. flexion + rotation left vs. flexion + rotation right) and knee angle (extended/stoop vs. flexed/squat) are investigated in randomized order.
  3. Functional tasks Three tests with two conditions in randomized order (exoskeleton: without vs. with) will be investigated in fixed order (stair-climbing; timed-up-and-go; course with various simulated industrial workstations).
  4. Angle-force relation Twelve conditions as combination of exoskeleton (without vs. with), knee angle (extended/stoop vs. flexed/squat) and trunk flexion angle (0 vs. 30 vs. 60 degrees) are investigated in randmized order.
Masking Description: Subjects and experimenters will not be blinded, because it will be obvious which task will be performed by the subjects and measurements need to be tracked by the experimenter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With exoskeleton, then without exoskeleton (Experimental): Subject will first perform the conditions (simulated, simplified, industrial standing work) with the exoskeleton, then without the exoskeleton.
  Interventions: Device: Laevo ®; Device: No Laevo ®
- Without exoskeleton, then with exoskeleton (Experimental): Subject will first perform the conditions (simulated, simplified, industrial standing work) without the exoskeleton, then with the exoskeleton.
  Interventions: Device: Laevo ®; Device: No Laevo ®

INTERVENTIONS:
Device: Laevo ® — A passive exoskeleton supporting the lower back during bending and lifting tasks (for more information, visit the manufacturer's website: http://en.laevo.nl/).
  Other Names: Exoskeleton
Device: No Laevo ® — The subjects will not wear any supporting device to perform the experiment, which serves as the control condition.
  Other Names: No exoskeleton

SUMMARY:
BACKGROUND Industrial tasks that are characterized by high loads, a high repetition rate, and/or awkward body postures, put employees at higher risk to develop work-related musculoskeletal disorders (WRMSD), especially low back pain. To counteract the prevalence of WRMSD, human-robot interaction could improve the power of a person and reduce the physical strain. For the lower back, a reduction of spinal loading could be helpful. The passive upper-extremity exoskeleton Laevo® is developed to support physically heavy work: it supports the back during bending and should, consequently, result in less low back pain (Laevo®, the Netherlands).

OBJECTIVES The primary aim of this study is to assess to what extent wearing the exoskeleton changes:

* muscular activity of the erector spinae and biceps femoris muscles;
* knee compression force;
* posture of the upper and lower spine, trunk, hips and knees; ...in different tasks (static vs. dynamic), different trunk postures (trunk flexion vs. trunk flexion and rotation) and different knee postures (straight vs. stooped).

Secondary aims of this study are to assess to what extent wearing the exoskeleton changes:

* muscular activity of the trapezius descendens, rectus abdominis, vastus medialis and gastrocnemius medialis;
* perceived discomfort;
* heart rate;
* internal loadings on the spine, using a lumbar spine model;
* the performance of subjects during functional activities (e.g., stair climbing) when wearing the exoskeleton (either turned on or off); ...in different tasks (static vs. dynamic), different trunk postures (trunk flexion vs. trunk flexion and rotation), different knee postures (stoop vs. squat), and different static holding positions(0° vs. 30° vs. 60°) with different weights (0kg vs. 8kg vs. 16kg).

DETAILED DESCRIPTION:
METHODS Different experiments will be performed.

1. The investigators will test six different experimental conditions in the laboratory, which are a combination of exoskeleton (with vs. without Laevo®), task (static vs. dynamic), and knee angle only for the dynamic task (flexed vs. extended). Within each combination, the investigators will test three different working directions (front vs. left vs. right), realized by changing the working posture (trunk flexion vs. left trunk rotation vs. right trunk rotation). Using the single Williams design for six conditions, the investigators estimated the sample size to include 36 subjects (i.e., a multiple of six). Using a force plate, acceleration and postural sensors, knee compression force can be estimated using 2D inverse modelling. With an electromyographic system, the muscle activity of selected target muscles at different body parts (i.e., legs, trunk, and shoulders) can be recorded. The heart rate will be recorded using electrocardiography.
2. The investigators will test four different conditions, which are a combination of exoskeleton (with vs. without Laevo®) and knee angle (flexed vs. extended). Within each combination, the investigators will test three different loads carried (0kg, 8kg, 16kg) and five different trunk flexion angles (0°, 30°, 60°, 60°, 30°). Muscle activity, position, heart rate and ground reaction forces will be recorded.
3. The investigators will test three different functional tests. The outcomes for this aim are time recorded for performing the functional or industrial task and perceived difficulty rated on an 11-point numeric rating scale.
4. The investigators will use the lumbar spine model developed by the research group Biomechanics and Biorobotics of the research cluster Simulation Technology of the University of Stuttgart. The model includes a detailed lumber spine with non-linear discs, ligaments, and muscles. Using the measurements of the experiment, this model is able to predict how internal forces in the lumbar spine change as a result of external forces (i.e., wearing and using the Laevo® exoskeleton).

ANALYSES Depending on the outcome parameter, different analyses will be performed including a various number of independent variables.

1. The effects of exoskeleton (with vs. without), task (static vs. dynamic), knee angle (flexed vs. extended; only for the dynamic task), and working posture (trunk flexion vs. left trunk rotation vs. right trunk rotation) will be assessed using a four-factor repeated-measures analysis of variance (RM-ANOVA) or a generalized estimating equation (GEE) which is more robust.
2. The effects of exoskeleton (with vs. without), knee angle (flexed vs. extended), load carried (0kg vs. 8kg vs. 16kg), and trunk flexion angle (0° vs. 30° vs. 60°) will be assessed using a RM-ANOVA or GEE.
3. The effect of exoskeleton (with vs. without) on time and perceived difficulty of each functional or industrial test will be assessed using a paired T-Test. In addition, the muscular load of several muscles will also be evaluated.

DATA PROTECTION All participating subjects will receive a refund of € 45 after study completion. Subjects will sign an informed consent and their data will be numerically pseudonymized to guarantee anonymity.

SIMULATED TASKS

1. Static sorting task, lasting 1.5 minutes, within which subjects are exposed to 6 experimental conditions: exoskeleton (2 levels: without vs. with) X working posture (3 levels: left trunk rotation vs. frontal orientation vs. right trunk rotation).
2. Dynamic lifting task, two sets of five repetitions each, within which subjects are exposed to 12 experimental conditons: exoskeleton (2 levels: without vs. with) X working posture (3 levels: left trunk rotation vs. frontal orientation vs. right trunk rotation) X knee angle (2 levels: extended/stoop vs. bent/squat).
3. Functional tasks: a course within which several occupationally relevant tasks (picking & placing, drilling) and standardized tests (sit-up-and-stand, stair walk) are evaluated on performance, subjectively perceived strain and muscle load.
4. Static holding task, for which subjects were exposed to 18 different conditions: exoskeleton (2 levels: without vs. with) X holding weight (3 levels: 0kg vs. 8kg vs. 16kg) X trunk flexion angle (3 levels: 0° vs. 30° vs. 60°).

IMPORTANT NOTE --- On this platform, results of the static sorting task ONLY will be reported. Results of other parts of the study will be reported in the respective publication. Links to these publications will be added as soon as they are published and available. --- IMPORTANT NOTE

ELIGIBILITY:
Inclusion Criteria:

* The participant will give his voluntary informed consent after receiving oral and written information of the content and goal of the study.

Exclusion Criteria:

* Aged <18 and >40 years;
* Female;
* BMI > 30 kg/m2;
* People under the influence of intoxicants, analgesics, or muscle relaxants;
* Alcohol abuse;
* People with cardiovascular diseases;
* People with a heart pacemaker;
* People with a disability who, due to their restriction at a workplace of this kind, will not be able to participate;
* People with Diabetes Mellitus;
* People with severe muscle contractions of the lower extremities, back or arms;
* People with acute ailments or pain;
* People who are unable to complete the examination program due to language or cognitive obstacles;
* Depending on the degree of severity, people with diseases of the veins and joints of the lower extremities, spine, muscle disorders, symptomatic neurological-psychiatric diseases, acute pain syndromes, maladies or other current diseases.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Occupational and Social Medicine and Health Services Research, University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Luger T, Bar M, Seibt R, Rieger MA, Steinhilber B. Using a Back Exoskeleton During Industrial and Functional Tasks-Effects on Muscle Activity, Posture, Performance, Usability, and Wearer Discomfort in a Laboratory Trial. Hum Factors. 2023 Feb;65(1):5-21. doi: 10.1177/00187208211007267. Epub 2021 Apr 16. PMID 33861139
- [Result] Luger T, Bar M, Seibt R, Rimmele P, Rieger MA, Steinhilber B. A passive back exoskeleton supporting symmetric and asymmetric lifting in stoop and squat posture reduces trunk and hip extensor muscle activity and adjusts body posture - A laboratory study. Appl Ergon. 2021 Nov;97:103530. doi: 10.1016/j.apergo.2021.103530. Epub 2021 Jul 16. PMID 34280658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteering participants were recruited via the collaborating investigators and by means of announcement e-mails to employees and students of the University and Hospital of Tübingen.
Pre-assignment Details: 39 volunteering participants were recruited, of which 2 were excluded from the study prior to the measurement due to a too high BMI (> 30 kg/m2). A 3rd participant was excluded because he was the first that was measured and we had to adjust a few things to the measurement afterwards.
Groups:
- First With Exoskeleton Then Without Exoskeleton: Subject will perform the conditions (simulated, simplified, industrial standing work) as described under "model description" first with and then without the exoskeleton.
- First Without Exoskeleton Then With Exoskelton: Subject will perform the conditions (simulated, simplified, industrial standing work) as described under "model description" first without and then with the exoskeleton.
Period: First Intervention
Arm/Group | First With Exoskeleton Then Without Exoskeleton | First Without Exoskeleton Then With Exoskelton
Started | 20 | 19
Completed | 19 | 17
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 1
Period: Second Intervention
Arm/Group | First With Exoskeleton Then Without Exoskeleton | First Without Exoskeleton Then With Exoskelton
Started | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: On the pre-measurement assessment, all volunteering participants were screened for eligability and basic information was collected, such as age.
Groups:
- With Exoskeleton, Then Without Exoskeleton: Subject first performed the conditions (simulated, simplified, industrial standing work) with the exoskeleton, then without the exoskeleton.
- Without Exoskeleton, Then With Exoskeleton: Subject first performed the conditions (simulated, simplified, industrial standing work) without the exoskeleton, then with the exoskeleton.
- Total: Total of all reporting groups
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (3.8) | 28.1 (4.6) | 25.9 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 19 | 17 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 17 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 19 | 17 | 36
Weight [Mean (Standard Deviation); unit: kg] | 73.3 (9.4) | 73.8 (8.5) | 73.5 (8.9)
Height [Mean (Standard Deviation); unit: cm] | 179.7 (6.3) | 178.0 (6.7) | 178.9 (6.4)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.6 (2.1) | 23.3 (2.1) | 22.9 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Muscular Activity of Erector Spinae Muscle.
Description: Root-mean-square (RMS) of the electrical activity of the erector spinae muscle using surface electromyography (sEMG). The sEMG signals will be continuously recorded, and the RMS will be normalized to a maximal voluntary contraction (%MVE) and averaged over the time period of each experimental condition.
Time Frame: Average RMS-value (%MVE) over the time period running from baseline (0 min) to directly after (1.5 min) the experimental condition
Population: The results of the effect of wearing the exoskeleton during the static task are reported below, without taking into account the working direction (frontal or lateral, i.e. without or with trunk rotation, respectively). Note: the overall number of participants analyzed deviates in the first arm because data of one subject was excluded.
Measure: Median (Inter-Quartile Range); unit: %MVE
Groups:
- With Exoskeleton, Then Without Exoskeleton: Subjects first performed the conditions (simulated, simplified, industrial standing work) with the exoskeleton, then without the exoskeleton.
- Without Exoskeleton, Then With Exoskeleton: Subjects first performed the conditions (simulated, simplified, industrial standing work) without the exoskeleton, then with the exoskeleton.
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton
Number analyzed (Participants) | 18 | 17
%MVE
  RMS-value during first intervention period | 11.2 [8.6 to 16.0] | 11.1 [8.6 to 14.8]
  RMS-value during second intervention period | 12.3 [9.0 to 17.6] | 10.4 [7.5 to 13.1]

2. Primary Outcome: Muscular Activity of Biceps Femoris Muscle.
Description: Root-mean-square (RMS) of the electrical activity of the biceps femoris muscle using surface electromyography (sEMG). The sEMG signals will be continuously recorded, and the RMS will be normalized to a reference voluntary contraction (%RVE) and averaged over the time period of each experimental condition.
Time Frame: Average RMS-value (%RVE) over the time period running from baseline (0 min) to directly after (1.5 min) the experimental condition
Population: The results of the effect of wearing the exoskeleton during the static task are reported below, without taking into account the working direction (frontal or lateral, i.e. without or with trunk rotation, respectively).
Measure: Median (Inter-Quartile Range); unit: %RVE
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton
Number analyzed (Participants) | 19 | 17
%RVE
  RMS during first intervention period | 26.6 [16.3 to 39.3] | 38.7 [23.9 to 57.5]
  RMS during second intervention period | 35.8 [24.4 to 45.8] | 31.3 [20.2 to 55.7]

3. Primary Outcome: Posture (Thoracic Kyphosis)
Description: The posture of the upper spine (thoracic kyphosis) determined using 2D gravimetric position sensors placed on the thoracic vertebrae T1 and lumbar vertebrae L1. The difference value between both sensors reflects the thoracic kyphosis, which was averaged over each experimental condition.
Time Frame: Average thoracic kyphosis over time period baseline (0 min) to directly after (1.5 min) the experimental condition
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton
Number analyzed (Participants) | 19 | 17
degrees
  Average angle during first intervention period | 12.0 [7.5 to 15.8] | 15.4 [8.0 to 21.0]
  Average angle during second intervention period | 14.5 [7.6 to 19.5] | 13.9 [8.8 to 21.3]

4. Primary Outcome: Posture (Lumbar Lordosis)
Description: The posture of the lower spine (lumbar lordosis) determined using 2D gravimetric position sensors placed on the lumbar vertebrae L1 and L5. The difference value between both sensors reflects the lumbar lordosis, which was averaged over each experimental condition.
Time Frame: Average lumbar lordosis over time period baseline (0 min) to directly after (1.5 min) the experimental condition
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton
Number analyzed (Participants) | 19 | 17
degrees
  Average angle during first intervention period | 11.8 [10.0 to 14.2] | 13.2 [9.4 to 17.7]
  Average angle during second intervention period | 12.2 [10.1 to 14.0] | 13.3 [10.4 to 16.1]

5. Primary Outcome: Posture (Trunk Flexion)
Description: The posture of the trunk determined using a 2D gravimetric position sensor placed on the thoracic vertebrae T10. The flexion angle of the sensor was averaged over each experimental condition.
Time Frame: Average trunk flexion over time period baseline (0 min) to directly after (1.5 min) the experimental condition
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton
Number analyzed (Participants) | 19 | 17
degrees
  Average angle during first intervention period | 38.5 [36.5 to 41.1] | 39.6 [35.6 to 42.2]
  Average angle during second intervention period | 37.9 [35.7 to 40.5] | 39.9 [35.9 to 43.5]

6. Primary Outcome: Posture (Hip Flexion)
Description: The posture of the hip (hip flexion) determined using 2D gravimetric position sensors placed on the lumbar vertebrae L5 and the upper leg (femur). The difference value between both sensors reflects the hip flexion, which was averaged over each experimental condition.
Time Frame: Average hip flexion over time period baseline (0 min) to directly after (1.5 min) the experimental condition
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton
Number analyzed (Participants) | 19 | 17
degrees
  Average angle during first intervention period | 39.9 [33.8 to 45.8] | 33.1 [24.7 to 38.4]
  Average angle during second intervention period | 29.8 [23.6 to 38.3] | 40.4 [32.1 to 47.1]

7. Primary Outcome: Posture (Knee Flexion)
Description: The posture of the knee (knee flexion) determined using 2D gravimetric position sensors placed on the upper leg (femur) and lower leg (tibia). The difference value between both sensors reflects the knee flexion, which was averaged over each experimental condition.
Time Frame: Average knee flexion over time period baseline (0 min) to directly after (1.5 min) the experimental condition
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton
Number analyzed (Participants) | 19 | 17
degrees
  Average angle during first intervention period | 16.4 [9.4 to 26.4] | 11.7 [3.7 to 17.5]
  Average angle during second intervention period | 9.0 [2.9 to 16.7] | 17.9 [10.5 to 25.6]

8. Primary Outcome: Knee Compression Force
Description: The knee compression force (KCF) is calculated using 2D inverse modelling with continuous recordings from 2D gravimetric position sensors (for joint angles) and a force plate (for ground reaction forces). The average knee compression force will be calculated over each experimental condition and summarized for both the left and right knee, since the task is executed in the frontal plane.
Time Frame: Average knee compression force (KCF) over the time period running from baseline (0 min) to directly after (1.5 min) the experimental condition
Population: For some of the participants, we could not analyze the knee compression force (KCF) data, because some information was missing to apply the modelling procedure.
Measure: Median (Inter-Quartile Range); unit: N
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton
Number analyzed (Participants) | 15 | 14
N
  Average KCF during first intervention period | 845 [741 to 897] | 742 [609 to 892]
  Average KCF during second intervention period | 807 [747 to 868] | 874 [660 to 963]

9. Secondary Outcome: Muscular Activity of Rectus Abdominis, Vastus Lateralis, Gastrocnemius Medialis and Trapezius Descendens Muscles.
Description: Root-mean-square (RMS) of the electrical activity of the rectus abdominis, vastus lateralis, gastrocnemius medialis and trapezius descendens muscles using surface electromyography (sEMG). The sEMG signals will be continuously recorded, and the RMS will be normalized to a refeernce voluntary contraction (%RVE) and averaged over the time period of each experimental condition.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: %RVE
Groups:
- Without Exoskeleton: Subjects performed the condition without the exoskeleton.
- With Exoskeleton: Subjects performed the condition with the exoskeleton.
Arm/Group | Without Exoskeleton | With Exoskeleton
Number analyzed (Participants) | 36 | 36
%RVE
  Rectus Abdominis | 1.85 [0.98 to 2.72] | 1.57 [0.88 to 2.26]
  Vastus Lateralis | 3.85 [2.06 to 5.64] | 3.35 [1.99 to 4.71]
  Gastrocnemius Medialis | 54.11 [30.63 to 77.59] | 54.11 [34.75 to 73.58]
  Trapezius Descendens | 3.77 [0.71 to 6.83] | 4.90 [1.21 to 8.60]

10. Secondary Outcome: Rating of Perceived Discomfort (RPD)
Description: Discomfort (RPD) was assessed using an 11-point numeric rating scale (NRS), ranging from 0 (no discomfort at all) to 10 (maximally imaginable discomfort). It was assessed directly before (0 min) and directly after (1.5 min) each experimental condition. The experimental conditions consisted of either static or dynamic tasks, that lasted up to 1.5 minutes.
Time Frame: Change from baseline (0 min) to directly after (1.5 min) both experimental conditions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | With Exoskeleton, Then Without Exoskeleton | Without Exoskeleton, Then With Exoskeleton
Number analyzed (Participants) | 19 | 17
units on a scale
  RPD after first intervention period | 0.3 (0.8) | 0.2 (0.6)
  RPD after second intervention period | 0.5 (1.0) | 0.2 (0.7)

11. Secondary Outcome: Heart Rate
Description: Continuous recording electrocardiography allows calculating the heart rate, a parameter reflecting the central stress state of the participant. The average heart rate will be calculated per time period.
Time Frame: Average heart activity over time period baseline (0 min) to directly after (1.5 min) the experimental condition
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Without Exoskeleton | With Exoskeleton
Number analyzed (Participants) | 36 | 36
beats per minute | 85.29 (10.19) | 83.16 (10.49)

12. Secondary Outcome: Evaluation of Workload
Description: The NASA Task Load Index (TLX) of Hart and Staveland (1988) will be used to evaluate workload. This standardized tool contains six dimensions (mental demand, physical demand, temporal demand, own performance, effort, frustration), of which each scale ranges from from 0 (low) to 100 (high).
  We will include three dimensions of interest, i.e. physical demand, temporal demand, effort, and calculate the unweighted average of the score of these three dimensions (Hoonakker et al. 2011).
Time Frame: Directly after the experimental condition during which the exoskeleton was worn (~ 4.5-6.5 min)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | With Exoskeleton | Without Exoskeleton
Number analyzed (Participants) | 36 | 36
units on a scale
  Physical Demand | 2.31 (1.58) | 1.67 (1.10)
  Temporal Demand | 1.10 (1.35) | 0.88 (1.01)
  Effort | 2.10 (1.30) | 1.49 (1.00)

13. Secondary Outcome: Self-developed Participant Evaluation Questionnaire
Description: This questionnaire will consist of questions about usability and acceptance of the intervention (the Laevo device), stemming from standardized questions from existing questionnaires, including:
  * the System Usability Scale (SUS): 10 statements about subjective perception of interaction with the Laevo system to be evaluated on a scale ranging from 1 (disagree) to 5 (agree);
  * the Technology Usage Inventory (TUI): 30 statements on technology-specific and psychological factors with respect to the Laevo to be evaluated on a scale ranging from 1 (not true) to 7 (true); of these 30 questions, the investigators include only 7 statements belonging to the domains 'usability' and 'skepticism'.
  The questionnaire can only be filled out after the condition within which the technology (here: exoskeleton) was used. That means that results are only provided and, thus, reported from the arm "with exoskeleton".
Time Frame: Directly after the experiment (~2.5 hours)
Population: Reportedin units on a scale:
  SUS: 0 (low usability) to 100 (high usability) TUI-userfriendliness: 3 (totaly not applicable) to 21 (totally applicable) TUI-scepticism: 4 (totaly not applicable) to 28 (totaly applicable)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | With Exoskeleton
Number analyzed (Participants) | 36
units on a scale
  System Usability Scale (SUS) - total score | 75.44 (12.87)
  Technology Usability Inventory (TUI) - user friendlines score | 17.92 (2.61)
  Technology Usability Inventory (TUI) - scepticims | 11.53 (4.08)

ADVERSE EVENTS:
Time Frame: One hour for each intervention.
Groups:
- With Exoskeleton: Subjects performed the conditions (simulated, simplified, industrial standing work) with the exoskeleton.
- Without Exoskeleton: Subjects performed the conditions (simulated, simplified, industrial standing work) without the exoskeleton.
Arm/Group | With Exoskeleton | Without Exoskeleton
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT03725982/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT03725982/ICF_001.pdf